CLINICAL TRIAL: NCT03194646
Title: An Open-label, Parallel-group, Randomized, Multicenter Study to Assess the Safety and Efficacy of Vilaprisan in Subjects With Uterine Fibroids Versus Standard of Care
Brief Title: Assess Safety and Efficacy of Vilaprisan in Subjects With Uterine Fibroids
Acronym: ASTEROID 6
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a change in the development program, the study was closed prematurely.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16953; 2016-004822-41 (EudraCT Number)
Record Dates: First submitted 2017-06-20; First posted 2017-06-21 (Actual); Results first posted 2021-08-26 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Uterine Fibroids
Keywords: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma | interventions — vilaprisan; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A1(3/1 regimen) (Experimental): 2.0 mg treatment of 12 weeks, each separated by 1 bleeding break
  Interventions: Drug: Vilaprisan (BAY1002670)
- A2(6/2 regimen) (Experimental): 2.0 mg treatment period of 24 weeks, each separated by 2 bleeding break
  Interventions: Drug: Vilaprisan (BAY1002670)
- A3(3/2 regimen) (Experimental): 2.0 mg treatment period of 12 weeks, each separated by 2 bleeding break
  Interventions: Drug: Vilaprisan (BAY1002670)
- B(Standard of care) (Other): Standard of care as determined by the investigators, this could be watch & wait or non-hormonal medical treatment
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — 2 mg of Vilaprisan once daily for 12 weeks, 4 treatment periods of 12 weeks, each separated by 1 bleeding episode (3/1 regimen).
  Arms: A1(3/1 regimen)
Drug: Vilaprisan (BAY1002670) — 2 mg of Vilaprisan once daily for 24 weeks, 2 treatment periods of 24 weeks, each separated by 2 bleeding episodes (6/2 regimen).
  Arms: A2(6/2 regimen)
Drug: Vilaprisan (BAY1002670) — 2 mg of Vilaprisan once daily for 12 weeks, 4 treatment periods of 12 weeks, each separated by 2 bleeding episodes (3/2 regimen).
  Arms: A3(3/2 regimen)
Other: Standard of care — Standard of care as determined by the investigators (including watch and wait, symptomatic nonhormonal)
  Arms: B(Standard of care)
Drug: Vilaprisan (BAY1002670) — 2 mg of Vilaprisan once daily for 12 weeks, 8 treatment periods of 12 weeks, each separated by 1 bleeding episode (3/1 regimen)
  Arms: A1(3/1 regimen)
Drug: Vilaprisan (BAY1002670) — 2 mg of Vilaprisan once daily for 24 weeks, 4 treatment periods of 24 weeks, each separated by 2 bleeding episodes (6/2 regimen)
  Arms: A2(6/2 regimen)
Drug: Vilaprisan (BAY1002670) — 2 mg of Vilaprisan once daily for 12 weeks, 6 treatment periods of 12 weeks, each separated by 2 bleeding episodes (3/2 regimen)
  Arms: A3(3/2 regimen)

SUMMARY:
The study was performed to assess the efficacy and safety of Vilaprisan in subjects with uterine fibroids compared to standard of care

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of uterine fibroid(s) documented by ultrasound at screening AND/OR during a uterine preserving procedure within 3 months prior to screening in subjects with high risk for recurrence
* At least one symptom of uterine fibroid(s) - bleeding, pelvic pressure/pain
* Good general health
* Normal or clinically insignificant cervical smear
* An endometrial biopsy performed during the screening period, without significant histological disorder
* Use of an acceptable nonhormonal method of contraception starting at Visit 1 until the end of the study

Exclusion Criteria:

* Pregnancy or lactation (less than 3 months since delivery, abortion, or lactation before start of treatment)
* Hypersensitivity to any ingredient of the study drug
* Any condition requiring immediate blood transfusion
* Any diseases, conditions, or medications that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Abuse of alcohol, drugs, or medicines (eg, laxatives)
* Use of other treatments that might interfere with the conduct of the study or the interpretation of the results
* Undiagnosed abnormal genital bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1272 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2024-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (219):
- United States (94):
  - Central Research Associates | Birmingham, AL, Birmingham, Alabama
  - Women's Health Alliance of Mobile, Mobile, Alabama
  - AMR - Mobile, AL, Mobile, Alabama
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences - Neurology, Little Rock, Arkansas
  - Diagnamics | Encinitas, CA, Encinitas, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - M3 Wake Research San Diego - Alvarado, San Diego, California
  - Women's Health Care Research | San Diego, CA, San Diego, California
  - West Coast OB/GYN Associates, San Diego, California
  - Advanced Women's Health Institute | Denver Office, Greenwood Village, CO, Greenwood Village, Colorado
  - Physicians' Research Options, LLC | Red Rocks OBGYN, Lakewood, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - IntimMedicine | Washington, DC, Washington D.C., District of Columbia
  - Helix Biomedics LLC | Boynton Beach, FL, Boynton Beach, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Doral Medical Research, Doral, Florida
  - M & O Clinical Research, LLC, Fort Lauderdale, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Axcess Medical Research, LLC, Loxahatchee Groves, Florida
  - Suncoast Clinical Research - Palm Harbor, Palm Harbor, Florida
  - ONCOVA Clinical Research, Inc., Saint Cloud, Florida
  - Swor Women's Care, Sarasota, Florida
  - Suncoast Clinical Research - New Port Richey, Trinity, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Atlanta Women's Research Institute, Inc. - Atlanta, Atlanta, Georgia
  - Medisense Inc at Atlantic Station, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Paramount Research Solutions | College Park Location, College Park, Georgia
  - Fellows Research Alliance, Inc | Savannah, GA, Savannah, Georgia
  - Journey Medical Research, Snellville, Georgia
  - Center For Women's Care, Palos Heights, Illinois
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Research Integrity, LLC, Owensboro, Kentucky
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Praetorian Pharmaceutical Research, LLC, Marrero, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Omni Fertility and Laser Institute, Shreveport, Louisiana
  - Johns Hopkins University School of Medicine, Columbia, Maryland
  - Baltimore Suburban Health, LLC, Pikesville, Maryland
  - Continental Clinical Solutions | Towson, MD, Towson, Maryland
  - Wayne State University Physicians Group, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Women's Clinic of Lincoln, P.C. | Lincoln, NE, Lincoln, Nebraska
  - M3 Wake Research - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Capital Health | Capital Health OBGYN Lawrenceville, Lawrenceville, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Bosque Women's Care | Albuquerque, NM, Albuquerque, New Mexico
  - SUNY Downstate Health Sciences University - Neurology, Brooklyn, New York
  - Integrated Medical Professionals, New York, New York
  - Columbia University Medical Center, New York, New York
  - Richmond ObGyn Associates PC, Staten Island, New York
  - Atrium Health Fertility Center, Charlotte, North Carolina
  - Carolina Women's Research & Wellness Center, Durham, North Carolina
  - Unified Women's Clinical Research - Greensboro, Greensboro, North Carolina
  - Unified Women's Clinical Research - Morehead City, Morehead City, North Carolina
  - Eastern Carolina Women's Center | New Bern, NC, New Bern, North Carolina
  - Women's Health Alliance, Raleigh, North Carolina
  - M3 Wake Research | Raleigh, NC, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Valaoras & Lewis OB/GYN, Winston-Salem, North Carolina
  - Clinical Inquest Center, Ltd., Beavercreek, Ohio
  - Miami Valley Hospital - Gynecology, Dayton, Ohio
  - HWC Women's Research Center | Englewood, OH, Englewood, Ohio
  - OHSU Hospital - Neurology, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center - Radiology, Hershey, Pennsylvania
  - Drexel University College of Medicine - Obstetrics and Gynecology, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania -, Philadelphia, Pennsylvania
  - Clinical Research Philadelphia | Philadelphia, PA, Philadelphia, Pennsylvania
  - MUSC Women's Health - Cannon St., Charleston, South Carolina
  - Vista Clinical Research, Columbia, South Carolina
  - VitaLink Research - Greenville, Greenville, South Carolina
  - Venus Gynecology, LLC | Myrtle Beach, SC, Myrtle Beach, South Carolina
  - Biocentric Health Resarch, West Columbia, South Carolina
  - ClinSearch, LLC, Hixson, Tennessee
  - Women's Physician Group, Memphis, Tennessee
  - Discovery Clinical Trials - Dallas, Dallas, Texas
  - Office of Dr. Delbert Alan Johns, MD, Fort Worth, Texas
  - Signature Gyn Services, Fort Worth, Texas
  - Advances in Health, INC. | Houston, TX, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - MacArthur Medical Center - OB/GYN, Irving, Texas
  - AdventHealth Family Medicine Clinic Lampasas, Lampasas, Texas
  - Willowbend Health and Wellness Associates, Plano, Texas
  - Seven Oaks Women's Center - Main Office - Medical Center, San Antonio, Texas
  - OB-GYN Physicians, Inc., Franklin, Virginia
  - Tidewater Clinical Research - Norfolk, Norfolk, Virginia
  - Virginia Physicians For Women, North Chesterfield, Virginia
  - Clinical Trials of Viriginia, Richmond, Virginia
  - Synexus Research, LLC, Richmond, Virginia
  - MultiCare Women's Health - Covington, Covington, Washington
- China (32):
  - Peking University First Hospital - Oncology Department, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Captial Medical University, Beijing, Beijing Municipality
  - 900th Hospital of Joint Logistics Support Force, Fuzhou, Fujian
  - Sun Yat-Sen Memorial Hosp. Sun Yat-Sen Univ., Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of TCM, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The 2nd Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Wuhan Tongji Reproductive Medicine Hospital, Wuhan, Hubei
  - Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu
  - NJ Drum Tower Hospital, the Affil Hos of NJ Univ Med School, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Second Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Second University Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - The Second Affliated Hospital of Wenzhou Medicial University, Wenzhou, Zhejiang
  - Beijing Hospital of Traditional Chinese Medicine, Beijing
  - Beijing Obstetrics and Gynecology Hospital,Capital Med.Uni., Beijing
  - Peking Union Medical College Hospital CAMS, Beijing
  - International Peace Maternity&Child Health Hospital of CWI, Shanghai
  - Changhai Hospital of Second Military Medical University, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - First Teaching Hosptial of Tianjin University of TCM, Tianjin
  - Tianjin Central Hospital of Gynecology obstetrics, Tianjin
- Czechia (8):
  - Centrum gynekologické rehabilitace, s.r.o., Písek, Jihoceský Kraj
  - Dr. Smrhova-Kovacs, Tábor, Jihočeský kraj
  - Fakultní nemocnice Brno, Brno
  - G-Centrum Olomouc s.r.o. Dr. Skrivanek, České Budějovice
  - Fakultní Nemocnice Hradec Kralové, Hradec Králové
  - MUDr. Radek Fiker s.r.o., Jihlava
  - Fakultní Nemocnice Olomouc, Olomouc
  - MUDr. Pavlina Nejedla s.r.o., Vodňany
- Finland (2):
  - Mehilainen | Mehilainen Kuopio, Kuopio
  - Lääkärikeskus Gyneko, Gynaecological Medical Center | Oulu, Finland, Oulu
- Queen Mary Hospital, Hong Kong, Hong Kong
- Japan (45):
  - Kano's Clinic for Women, Nagoya, Aichi-ken
  - Kyoritsu Narashinodai Hospital, Funabashi, Chiba
  - Juno Vesta Clinic Hatta, Matsudo, Chiba
  - Aso Iizuka Hospital, Iizuka, Fukuoka
  - Jusendo Geneal Hospital Yuasa Foundation, Kōriyama, Fukushima
  - Sato Hospital, Takasaki, Gunma
  - Primo Women's Clinic, Ebetsu, Hokkaido
  - Sapporo Maternity Women's Hospital, Sapporo, Hokkaido
  - Sapporo Shiroishi Obstetrics and Gynecology Hospital, Sapporo, Hokkaido
  - Hashimoto Clinic, Sapporo, Hokkaido
  - Ena Odori Clinic, Sapporo, Hokkaido
  - Sapporo Maternity Women's Minami1jo Clinic, Sapporo, Hokkaido
  - SAPPORO MEDICAL CENTER, NTT East Corporation, Sapporo, Hokkaido
  - Sapporo West Ladies Clinic, Sapporo, Hokkaido
  - Yoshio Clinic, Sapporo, Hokkaido
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Asahi-Clinic, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Second Kawasaki Saiwai Clinic, Kawasaki, Kanagawa
  - Kurashiki Medical Clinic, Kurashiki, Okayama-ken
  - Suita Municipal Hospital, Suita, Osaka
  - Medical Topia Soka Hospital, Sōka, Saitama
  - Fuyo Association Seirei Numazu Hospital, Numazu, Shizuoka
  - Sei Womens Clinic, Bunkyo, Tokyo
  - Ginza Yoshida Clinic, Chuo-ku, Tokyo
  - Women's wellness Tsushima Ruriko josei life clinic Ginza, Chuo-ku, Tokyo
  - St.Luke's International Hospital, Chuoku, Tokyo
  - Akazawa Clinic, Fuchū, Tokyo
  - Medical Corp. Seikoukai New Medical Research System Clinic, Hachiōji, Tokyo
  - Toranomon Womens Clinic, Minato, Tokyo
  - Akasakamitsuke Miyazaki Obstetrics and Gynecology Clinic, Minato, Tokyo
  - Shirokane Ladies' Clinic, Minato, Tokyo
  - Yokokura Clinic, Minato-ku, Tokyo
  - Kugayama Hospital, Setagaya-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Ikebukuro Metropolitan Clinic, Toshima-ku, Tokyo
  - Kato Internal medicine and Gynecology Clinic, Fukui
  - Sano Wemen's Clinic, Fukuoka
  - Unoki Clinic, Kagoshima
  - Medical corporation keizukai Chayamachi Ladies Clinic, Osaka
  - Chayamachi ladies Clinic Hommachi, Osaka
  - Medical Corporation Koshinkai Nomura Clinic Namba, Osaka
  - Izuma Clinic, Osaka
  - Shizuoka Saiseikai General Hospital, Shizuoka
  - Shizuoka City Shimizu Hospital, Shizuoka
- Mexico (3):
  - Hospital Universitario "José Eleuterio González", Monterrey, Nuevo León
  - Centro Integral Médico de San Juan del Río S. C., San Juan del Río, Querétaro
  - Sanatorio Alcocer Pozo S. A. de C. V., Querétaro
- Norway (3):
  - Kirkeparken Spesialistpraksis, Fredrikstad
  - Nesttun Spesialistpraksis AS, Nesttun
  - Medicus AS, Trondheim
- Poland (7):
  - Prywatna Klinika Ginekologiczno-Poloznicza, Bialystok
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Gyncentrum Sp. z o.o., Katowice
  - Prywatny Gabinet Lekarski Ginekologia, Poloznictwo i Ultr., Lodz
  - Centrum Medyczne Chodzki, Lublin
  - Specjalistyczny Gabinet Ginekologiczno-Polozniczy, Lublin
- Russia (9):
  - Scientific Center of family health & human reprod. problems, Irkutsk
  - Regional Clinical Hospital #2, Krasnodar
  - Krasnoyarsk regional perinatal center, Krasnoyarsk
  - City Clinical Hospital #13 Moscow, Moscow
  - Endocrinology Research Center, Moscow
  - St. Petersburg Medical University n.a. I.P. Pavlov, Saint Petersburg
  - Granti-Med, Saint Petersburg
  - Scien. Res. Institute of Obsterics, Gyn. & Reproduction, Saint Petersburg
  - Close Joint Stock Company "Medical Company IDK", Samara
- South Africa (7):
  - Dr L Reynders Practice, Lyttelton Manor, Gauteng
  - University of Pretoria, Clinical Research Unit, Pretoria, Gauteng
  - Femway Inc, Umhlanga, KwaZulu-Natal
  - Durban International Clinical Research Site, Wentworth, KwaZulu-Natal
  - Drs AEVITAS Clinic (Pty) Ltd, Cape Town, Western Cape
  - University of Cape Town Clinical Research Centre, Cape Town, Western Cape
  - Clintrials Centre for Clinical Research, Panorama, Western Cape
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Mahidol, Bangkok
- Turkey (Türkiye) (6):
  - Cukurova Universitesi Tip Fakultesi Hastanesi, Adana
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Etlik Zubeyde Hanim Kadin Hastaliklari Egitim Arastirma Hast, Ankara
  - Uludag Universitesi Tip Fakultesi, Bursa
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Istanbul Universitesi Cerrahpasa-Cerrahpasa Tip Fakultesi, Istanbul

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 219 study centers in 13 countries worldwide between 30-Jun-2017 (first participant first visit) and 11-Jul-2024 (last participant last visit).
Pre-assignment Details: Overall, 2368 participants were screened. Of the 2368 screened participants, 1096 (46.3%) participants were not randomized to treatment due to screen failures. 1272 (53.7%) participants were randomized and 1238 (52.3%) participants received study treatment.
Groups:
- Vilaprisan 2 mg A1 (3/1 Regimen): 4 treatment periods of 12 weeks, each separated by 1 bleeding episode
- Vilaprisan 2 mg A2 (6/2 Regimen): 2 treatment periods of 24 weeks, separated by 2 bleeding episodes
- Vilaprisan 2 mg A3 (3/2 Regimen): 3 treatment periods of 12 weeks, each separated by 2 bleeding episodes
- B (Standard of Care): Standard of care symptomatic nonhormonal medical treatment as determined by the investigators and/or watch and wait
Period: Overall Study
Arm/Group | Vilaprisan 2 mg A1 (3/1 Regimen) | Vilaprisan 2 mg A2 (6/2 Regimen) | Vilaprisan 2 mg A3 (3/2 Regimen) | B (Standard of Care)
Started (Randomized) | 363 | 361 | 183 | 365
Treated (Treated (with study drug or study drug administration status unknown or randomized to Standard of Care)) | 349 | 347 | 177 | 365
Completed | 59 | 93 | 44 | 85
Not Completed | 304 | 268 | 139 | 280
Not completed — Adverse Event | 24 | 25 | 14 | 17
Not completed — Lack of Efficacy | 4 | 2 | 2 | 12
Not completed — Lost to Follow-up | 30 | 22 | 12 | 35
Not completed — Non-compliance with study drug | 4 | 0 | 1 | 1
Not completed — Other | 89 | 68 | 34 | 31
Not completed — Physician Decision | 7 | 9 | 5 | 4
Not completed — Pregnancy | 4 | 5 | 1 | 2
Not completed — Protocol Violation | 4 | 2 | 1 | 1
Not completed — Site terminated by sponsor | 0 | 0 | 2 | 0
Not completed — Study terminated by sponsor | 62 | 61 | 30 | 34
Not completed — Withdrawal by Subject | 75 | 74 | 36 | 131
Not completed — Missing | 1 | 0 | 1 | 12

BASELINE CHARACTERISTICS:
Population: Participants in Full analysis set (FAS) was analyzed. The FAS consisted of all randomized subjects, excluding randomized subjects who did not start treatment Period 1 (never received study drug) due to the study being temporarily paused, including 1264 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vilaprisan 2 mg A1 (3/1 Regimen) | Vilaprisan 2 mg A2 (6/2 Regimen) | Vilaprisan 2 mg A3 (3/2 Regimen) | B (Standard of Care) | Total
Number analyzed (Participants) | 361 | 357 | 181 | 365 | 1264
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.7 (5.9) | 41.6 (6.0) | 41.9 (6.0) | 42.2 (6.1) | 41.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 361 | 357 | 181 | 365 | 1264
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 36 | 15 | 35 | 114
  Not Hispanic or Latino | 330 | 319 | 166 | 327 | 1142
  Unknown or Not Reported | 3 | 2 | 0 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 2 | 3 | 17
  Asian | 124 | 126 | 64 | 129 | 443
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 99 | 90 | 43 | 100 | 332
  White | 129 | 129 | 71 | 132 | 461
  More than one race | 3 | 3 | 0 | 0 | 6
  Unknown or Not Reported | 0 | 3 | 1 | 1 | 5
Baseline bone mineral density (BMD) of lumbar spine, hip and femoral neck [Mean (Standard Deviation); unit: g/cm^2] — The baseline data of BMD measured by dual-energy X-ray absorptiometry (DEXA) scan for lumbar spine, hip and femoral neck is provided in below table. Population: Safety analysis set (SAF) was analyzed. SAF: All participants randomized to vilaprisan treatment groups who took at least 1 dose of study drug and all participants randomized to group B (standard of care) treatment group were included in the SAF. Participants were analyzed as treated. Some data in baseline was missing.
  g/cm^2
    Lumbar spine: number analyzed (Participants) | 339 | 338 | 174 | 350 | 1201
    Lumbar spine | 1.1468 (0.1869) | 1.1653 (0.1889) | 1.1560 (0.1807) | 1.1532 (0.1851) | 1.1552 (0.1860)
    Hip: number analyzed (Participants) | 340 | 337 | 174 | 357 | 1208
    Hip | 0.9998 (0.1528) | 1.0044 (0.1614) | 1.0063 (0.1508) | 0.9944 (0.1486) | 1.0004 (0.1536)
    Femoral neck: number analyzed (Participants) | 340 | 337 | 174 | 357 | 1208
    Femoral neck | 0.9050 (0.1700) | 0.9174 (0.1808) | 0.9150 (0.1730) | 0.9021 (0.1703) | 0.9090 (0.1735)
Endometrial thickness [Mean (Standard Deviation); unit: Millimeters] — Ultrasound examinations were performed. Endometrial thickness was measured in the medio-sagittal section as double-layer in millimeters. Baseline data (Last non-missing value before reference start date) of endometrial thickness is provided in below table. Population: Safety analysis set (SAF) was analyzed. SAF: All participants randomized to vilaprisan treatment groups who took at least 1 dose of study drug and all participants randomized to group B (standard of care) treatment group were included in the SAF. Participants were analyzed as treated. Some data in baseline were missing.
  Millimeters
    number analyzed (Participants) | 348 | 344 | 176 | 363 | 1231
    (all) | 8.3 (3.8) | 8.3 (4.0) | 8.6 (3.8) | 8.7 (4.3) | 8.5 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Bone Mineral Density (BMD) of Lumbar Spine
Description: The percentage change in BMD (measured by dual-energy X-ray absorptiometry (DEXA) scan) of lumbar spine from baseline to about one year after start of treatment (SoT) in all randomized and treated participants with measurements at those 2 time points in each treatment group.
Time Frame: From baseline to about 1 year after start of treatment
Population: Safety analysis set (SAF) was analyzed. SAF: All participants randomized to vilaprisan treatment groups who took at least 1 dose of study drug and all participants randomized to group B (standard of care) treatment group were included in the SAF. Participants were analyzed as treated. Overall number of participants analyzed represents number of participants without missing data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Vilaprisan 2 mg A1 (3/1 Regimen) | Vilaprisan 2 mg A2 (6/2 Regimen) | Vilaprisan 2 mg A3 (3/2 Regimen) | B (Standard of Care)
Number analyzed (Participants) | 112 | 143 | 57 | 181
Percentage change | -1.56 (2.72) | -2.04 (2.50) | -1.51 (2.28) | 0.29 (2.36)
Statistical Analysis 1: Comparison: Vilaprisan 2 mg A1 (3/1 Regimen) vs B (Standard of Care); Test type: Other; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-2.44 to -1.26]
Statistical Analysis 2: Comparison: Vilaprisan 2 mg A2 (6/2 Regimen) vs B (Standard of Care); Test type: Other; Mean Difference (Final Values) = -2.34, 95% CI 2-sided [-2.87 to -1.80]
Statistical Analysis 3: Comparison: Vilaprisan 2 mg A3 (3/2 Regimen) vs B (Standard of Care); Test type: Other; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-2.51 to -1.10]

2. Secondary Outcome: Number of Bleeding Days
Description: Number of bleeding days were defined from Day 1 of the first treatment period until the day before a new treatment period would start again following the last treatment period for that respective treatment group. Number to be normalized by 28 days
Time Frame: Treatment phase: approximately 1 year
Population: FAS was analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Vilaprisan 2 mg A1 (3/1 Regimen) | Vilaprisan 2 mg A2 (6/2 Regimen) | Vilaprisan 2 mg A3 (3/2 Regimen) | B (Standard of Care)
Number analyzed (Participants) | 349 | 347 | 177 | 365
Days | 1.57 (1.99) | 1.74 (2.52) | 1.81 (1.24) | 4.72 (4.60)

3. Secondary Outcome: Number of Participants With Endometrial Histology Findings by Endometrial Biopsy Main Results (Majority Read, Main Diagnosis)
Description: Number of participants with endometrial histology findings, e.g. benign endometrium, presence or absence of hyperplasia or malignancy
Time Frame: Up to 3 years (from study treatment start to end of study)
Population: SAF was analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Vilaprisan 2 mg A1 (3/1 Regimen): 4 treatment periods of 12 weeks, each separated by 1 bleeding episode (3/1 regimen)
Arm/Group | Vilaprisan 2 mg A1 (3/1 Regimen) | Vilaprisan 2 mg A2 (6/2 Regimen) | Vilaprisan 2 mg A3 (3/2 Regimen) | B (Standard of Care)
Number analyzed (Participants) | 349 | 347 | 177 | 365
Participants
  Adequate endometrial tissue: number analyzed (Participants) | 349 | 347 | 177 | 364
  Adequate endometrial tissue | 346 | 346 | 175 | 359
  Benign Endometrium: number analyzed (Participants) | 346 | 346 | 175 | 359
  Benign Endometrium | 346 | 346 | 175 | 359
  Hyperplasia WHO 2014, no atypia: number analyzed (Participants) | 346 | 346 | 175 | 359
  Hyperplasia WHO 2014, no atypia | 0 | 0 | 0 | 0
  Hyperplasia WHO 2014, atypia: number analyzed (Participants) | 346 | 346 | 175 | 359
  Hyperplasia WHO 2014, atypia | 0 | 0 | 0 | 0
  Malignant Neoplasm: number analyzed (Participants) | 346 | 346 | 175 | 359
  Malignant Neoplasm | 0 | 0 | 0 | 0
  Endometrial Polyps: number analyzed (Participants) | 346 | 346 | 175 | 359
  Endometrial Polyps | 6 | 8 | 4 | 4

4. Secondary Outcome: Change From Baseline in Endometrial Thickness
Description: Ultrasound examinations were performed. Endometrial thickness was measured in the medio-sagittal section as double-layer in millimeters. Summary statistics for change from baseline (worst measurement during baseline period) in endometrial thickness was provided in below table.
Time Frame: Treatment phase: approximately 1 year, follow-up phase: up to 2 years
Population: SAF was analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Vilaprisan 2 mg A1 (3/1 Regimen) | Vilaprisan 2 mg A2 (6/2 Regimen) | Vilaprisan 2 mg A3 (3/2 Regimen) | B (Standard of Care)
Number analyzed (Participants) | 349 | 347 | 177 | 365
Millimeters
  Baseline: number analyzed (Participants) | 348 | 344 | 176 | 363
  Baseline | 10.4 (4.0) | 10.7 (4.0) | 10.9 (4.0) | 11.0 (4.4)
  Treatment phase (change from baseline): number analyzed (Participants) | 264 | 318 | 127 | 316
  Treatment phase (change from baseline) | -0.5 (5.6) | -0.2 (5.7) | -0.9 (4.7) | -0.4 (4.5)
  Follow up phase (change from baseline): number analyzed (Participants) | 323 | 307 | 163 | 142
  Follow up phase (change from baseline) | -0.2 (5.2) | -0.3 (5.7) | -1.1 (4.5) | -2.7 (4.6)

5. Secondary Outcome: Percentage Change From Baseline in BMD Measured at Lumbar Spine (Other Time Points Not Mentioned as Primary Safety Variable) and Hip/Femoral Neck
Description: Percentage change in BMD (measured by dual-energy X-ray absorptiometry (DEXA) scan) of lumbar spine (other time points not mentioned as primary safety analysis), hip, and femoral neck from baseline was analyzed using the same statistical methods as used for the primary variable.
Time Frame: Treatment phase: approximately 1 year, follow-up phase: up to 2 years
Population: SAF was analyzed. Percentage change from baseline in BMD of lumbar spine, hip and femoral neck was presented by time interval in below table.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Vilaprisan 2 mg A1 (3/1 Regimen) | Vilaprisan 2 mg A2 (6/2 Regimen) | Vilaprisan 2 mg A3 (3/2 Regimen) | B (Standard of Care)
Number analyzed (Participants) | 349 | 347 | 177 | 365
Percentage change
  Lumbar spine - Month 6 on treatment: number analyzed (Participants) | 15 | 35 | 8 | 8
  Lumbar spine - Month 6 on treatment | -0.18 (1.70) | -0.49 (2.74) | 0.51 (2.52) | -0.88 (2.60)
  Lumbar spine - End of treatment: number analyzed (Participants) | 100 | 172 | 67 | 161
  Lumbar spine - End of treatment | -1.48 (2.68) | -1.76 (2.64) | -1.22 (2.36) | 0.13 (2.38)
  Lumbar spine - Month 6 post treatment: number analyzed (Participants) | 127 | 144 | 75 | 93
  Lumbar spine - Month 6 post treatment | -0.69 (3.30) | -0.89 (2.72) | -0.57 (2.36) | -0.17 (2.76)
  Lumbar spine - Month 12 post treatment: number analyzed (Participants) | 7 | 13 | 6 | 13
  Lumbar spine - Month 12 post treatment | -0.10 (2.81) | -0.45 (3.61) | 0.86 (2.73) | 1.03 (6.79)
  Lumbar spine - End of follow up: number analyzed (Participants) | 246 | 245 | 125 | 113
  Lumbar spine - End of follow up | -0.64 (4.23) | -0.28 (4.11) | -0.38 (4.26) | -0.07 (3.49)
  Hip - Month 6 on treatment: number analyzed (Participants) | 16 | 35 | 8 | 8
  Hip - Month 6 on treatment | -1.00 (2.89) | -0.48 (2.49) | 1.54 (1.21) | -0.23 (1.81)
  Hip - Month 12 on treatment: number analyzed (Participants) | 112 | 143 | 56 | 182
  Hip - Month 12 on treatment | -0.84 (2.19) | -0.99 (2.23) | -0.91 (2.68) | -0.03 (2.47)
  Hip - End of treatment: number analyzed (Participants) | 101 | 172 | 67 | 162
  Hip - End of treatment | -0.85 (2.28) | -0.91 (2.34) | -0.61 (2.63) | -0.06 (2.65)
  Hip - Month 6 post treatment: number analyzed (Participants) | 127 | 144 | 74 | 93
  Hip - Month 6 post treatment | -0.45 (2.30) | -0.62 (2.60) | -0.54 (3.06) | 0.20 (2.72)
  Hip - Month 12 post treatment: number analyzed (Participants) | 7 | 13 | 6 | 14
  Hip - Month 12 post treatment | -0.72 (1.95) | -0.33 (1.91) | 1.41 (2.22) | -0.23 (3.77)
  Hip - End of follow up: number analyzed (Participants) | 247 | 244 | 125 | 114
  Hip - End of follow up | -0.80 (3.06) | -0.03 (3.85) | -0.20 (3.81) | 0.08 (2.91)
  Femoral neck - Month 6 on treatment: number analyzed (Participants) | 16 | 35 | 8 | 8
  Femoral neck - Month 6 on treatment | -0.71 (2.69) | 0.66 (3.27) | 1.23 (3.08) | 0.08 (3.80)
  Femoral neck - Month 12 on treatment: number analyzed (Participants) | 112 | 143 | 56 | 182
  Femoral neck - Month 12 on treatment | -0.84 (3.42) | -0.64 (3.45) | -0.66 (3.07) | -0.01 (3.42)
  Femoral neck - End of treatment: number analyzed (Participants) | 101 | 172 | 67 | 162
  Femoral neck - End of treatment | -1.12 (3.37) | -0.36 (3.46) | -0.42 (3.21) | -0.02 (3.47)
  Femoral neck - Month 6 post treatment: number analyzed (Participants) | 127 | 144 | 74 | 93
  Femoral neck - Month 6 post treatment | -0.87 (3.45) | -0.49 (3.52) | -0.35 (3.80) | -0.42 (3.32)
  Femoral neck - Month 12 post treatment: number analyzed (Participants) | 7 | 13 | 6 | 14
  Femoral neck - Month 12 post treatment | -0.82 (3.83) | -1.27 (3.60) | -0.65 (1.06) | 1.40 (5.19)
  Femoral neck - End of follow up: number analyzed (Participants) | 247 | 244 | 125 | 114
  Femoral neck - End of follow up | -0.90 (4.41) | -0.09 (5.16) | -0.52 (5.70) | -0.34 (3.73)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs): From first application of study medication up to 60 calendar days after end of study medication intake (mean duration 321 days). Post-treatment AEs: All AEs that started from Day 61 after end of study medication intake (mean duration 314 days for all participants until premature termination of the study, and 1572 days for Turkish participants who continued follow-up up to 5 years after individual end of study medication intake unless they withdrew).
Groups:
- Vilaprisan 2 mg A1 (3/1 Regimen) - Treatment Emergent AEs; Vilaprisan 2 mg A1 (3/1 Regimen) - Post Treatment AEs: 4 treatment periods of 12 weeks, each separated by 1 bleeding episode (3/1 regimen)
- Vilaprisan 2 mg A2 (6/2 Regimen) - Treatment Emergent AEs; Vilaprisan 2 mg A2 (6/2 Regimen) - Post Treatment AEs: 2 treatment periods of 24 weeks, separated by 2 bleeding episodes
- Vilaprisan 2 mg A3 (3/2 Regimen) - Treatment Emergent AEs; Vilaprisan 2 mg A3 (3/2 Regimen) - Post Treatment AEs: 3 treatment periods of 12 weeks, each separated by 2 bleeding episodes
- Standard of Care B - Treatment Emergent AEs; Standard of Care B - Post Treatment AEs: Standard of care symptomatic nonhormonal medical treatment as determined by the investigators and/or watch and wait
Arm/Group | Vilaprisan 2 mg A1 (3/1 Regimen) - Treatment Emergent AEs | Vilaprisan 2 mg A2 (6/2 Regimen) - Treatment Emergent AEs | Vilaprisan 2 mg A3 (3/2 Regimen) - Treatment Emergent AEs | Standard of Care B - Treatment Emergent AEs | Vilaprisan 2 mg A1 (3/1 Regimen) - Post Treatment AEs | Vilaprisan 2 mg A2 (6/2 Regimen) - Post Treatment AEs | Vilaprisan 2 mg A3 (3/2 Regimen) - Post Treatment AEs | Standard of Care B - Post Treatment AEs
All-Cause Mortality (participants affected / at risk) | 0/349 | 0/347 | 0/177 | 0/365 | 0/349 | 0/347 | 0/177 | 0/365
Serious Adverse Events (participants affected / at risk) | 15/349 | 17/347 | 6/177 | 17/365 | 54/349 | 42/347 | 27/177 | 7/365
Other Adverse Events (participants affected / at risk) | 136/349 | 152/347 | 56/177 | 90/365 | 75/349 | 67/347 | 44/177 | 14/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilaprisan 2 mg A1 (3/1 Regimen) - Treatment Emergent AEs (N=349) | Vilaprisan 2 mg A2 (6/2 Regimen) - Treatment Emergent AEs (N=347) | Vilaprisan 2 mg A3 (3/2 Regimen) - Treatment Emergent AEs (N=177) | Standard of Care B - Treatment Emergent AEs (N=365) | Vilaprisan 2 mg A1 (3/1 Regimen) - Post Treatment AEs (N=349) | Vilaprisan 2 mg A2 (6/2 Regimen) - Post Treatment AEs (N=347) | Vilaprisan 2 mg A3 (3/2 Regimen) - Post Treatment AEs (N=177) | Standard of Care B - Post Treatment AEs (N=365)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous angioma of brain (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRCA1 gene mutation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Primary hyperaldosteronism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biopsy peritoneum (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Norepinephrine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scan adrenal gland abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 2 (2) | 2 (2) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 5 (5) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine myoma expulsion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal epidural haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pelvic adhesions (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 17 (17) | 15 (15) | 8 (8) | 1 (1)
Mastectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myomectomy (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 6 (6) | 4 (4) | 2 (2) | 1 (1)
Salpingectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Simple mastectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Endometrial ablation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyst removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal adhesion lysis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hysterosalpingectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Meniscus removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine dilation and curettage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma embolisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous angioma of brain (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRCA1 gene mutation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Primary hyperaldosteronism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biopsy peritoneum (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Norepinephrine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scan adrenal gland abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 2 (2) | 2 (2) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 5 (5) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Degeneration of uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine myoma expulsion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal epidural haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pelvic adhesions (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic organ prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia with cellular atypia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 18 (18) | 16 (16) | 8 (8) | 1 (1)
Mastectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myomectomy (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 6 (6) | 5 (5) | 2 (2) | 1 (1)
Salpingectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Simple mastectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Endometrial ablation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyst removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hysterosalpingectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Meniscus removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine dilation and curettage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine artery embolisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal adhesiolysis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilaprisan 2 mg A1 (3/1 Regimen) - Treatment Emergent AEs (N=349) | Vilaprisan 2 mg A2 (6/2 Regimen) - Treatment Emergent AEs (N=347) | Vilaprisan 2 mg A3 (3/2 Regimen) - Treatment Emergent AEs (N=177) | Standard of Care B - Treatment Emergent AEs (N=365) | Vilaprisan 2 mg A1 (3/1 Regimen) - Post Treatment AEs (N=349) | Vilaprisan 2 mg A2 (6/2 Regimen) - Post Treatment AEs (N=347) | Vilaprisan 2 mg A3 (3/2 Regimen) - Post Treatment AEs (N=177) | Standard of Care B - Post Treatment AEs (N=365)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 8 (8) | 3 (3) | 29 (30) | 10 (10) | 12 (12) | 8 (8) | 1 (1)
Fatigue (General disorders) | 13 (13) | 20 (20) | 6 (6) | 18 (20) | 2 (2) | 3 (3) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 37 (51) | 42 (55) | 14 (15) | 12 (16) | 14 (22) | 12 (16) | 4 (4) | 0 (0)
Bone density decreased (Investigations) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 27 (27) | 25 (25) | 15 (15) | 6 (6)
Headache (Nervous system disorders) | 30 (43) | 24 (37) | 9 (9) | 7 (13) | 6 (6) | 2 (2) | 4 (4) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 16 (26) | 24 (45) | 9 (15) | 6 (8) | 16 (34) | 10 (15) | 2 (2) | 3 (3)
Endometrial thickening (Reproductive system and breast disorders) | 28 (34) | 39 (44) | 9 (9) | 13 (16) | 2 (3) | 4 (4) | 7 (7) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 12 (13) | 10 (10) | 3 (3) | 27 (30) | 16 (21) | 6 (8) | 8 (9) | 1 (1)
Hot flush (Vascular disorders) | 40 (53) | 44 (51) | 20 (24) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 8 (8) | 3 (3) | 29 (30) | 10 (10) | 12 (12) | 8 (8) | 1 (1)
Fatigue (General disorders) | 13 (13) | 20 (20) | 6 (6) | 18 (20) | 2 (2) | 3 (3) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 37 (51) | 42 (55) | 14 (15) | 12 (16) | 14 (22) | 12 (16) | 4 (4) | 0 (0)
Bone density decreased (Investigations) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 27 (27) | 25 (25) | 15 (15) | 6 (6)
Headache (Nervous system disorders) | 30 (43) | 24 (37) | 9 (9) | 7 (13) | 6 (6) | 2 (2) | 4 (4) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 16 (26) | 24 (45) | 9 (15) | 6 (8) | 16 (34) | 10 (15) | 2 (2) | 3 (3)
Endometrial thickening (Reproductive system and breast disorders) | 28 (34) | 39 (44) | 9 (9) | 13 (16) | 2 (3) | 4 (4) | 7 (7) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 12 (13) | 10 (10) | 3 (3) | 27 (30) | 16 (21) | 6 (8) | 8 (9) | 1 (1)
Hot flush (Vascular disorders) | 40 (53) | 44 (51) | 20 (24) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was ended prematurely. On top of the data included in the previous summary of results after primary completion, this final summary of results adds adverse event data from long term follow-up of subjects in Turkey as per local requirements. This was to ensure follow-up of all Turkish subjects for 5 years after end of study medication intake.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03194646/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT03194646/SAP_001.pdf